CLINICAL TRIAL: NCT05932095
Title: TCM Daoyin in the Treatment of Patients With Anxiety State: A Pilot Study
Brief Title: TCM Daoyin in the Treatment of Patients With Anxiety State
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Lu Ying, MM, assistant researcher, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ZY(2021-2023)- 0105-07
Record Dates: First submitted 2023-06-11; First posted 2023-07-06 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Anxiety State
Keywords: TCM Daoyin; Anxiety; Randomized controlled trial
MeSH Terms: conditions — Anxiety Disorders | interventions — Qigong

STUDY DESIGN:
Intervention Model Description: This is a 12-week, randomized controlled trial with an additional healthy control group. Patients with anxiety state are randomized 1:1 to either the TCM Daoyin intervention group or the health education control group (10 participants each). Additionally, 10 healthy volunteers will be enrolled as a non-randomized healthy control group for data comparison.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors were blinded to the group allocation of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TCM Daoyin intervention group (Experimental): Participants randomized to TCM Daoyin intervention group receive health education plus a TCM Daoyin training program. The TCM Daoyin training program was a 12-week, instructor-led group training program.
  Interventions: Behavioral: TCM Daoyin; Behavioral: Health education
- Health education control group (Active Comparator): Participants randomized to the health education control group only receive health education and no additional training program.
  Interventions: Behavioral: Health education
- Healthy Control (No Intervention): Healthy volunteers for data comparison, receiving no intervention.

INTERVENTIONS:
Behavioral: TCM Daoyin — The TCM Daoyin training program consisted of two 90-min training classes and at least five 30-min at-home practice sessions per week for 12-weeks. All sessions included 10 min of warmup and 10 min of cooldown.
  Other Names: Qigong
  Arms: TCM Daoyin intervention group
Behavioral: Health education — Health education is provided by psychologist and TCM doctor, including work, rest, diet and other basic programs.
  Arms: Health education control group; TCM Daoyin intervention group

SUMMARY:
In recent years, the number of people with symptoms of anxiety are on the rise. TCM Daoyin is a promising intervention for anxiety. This study is designed to allow researchers to better understand the changes in anxiety symptom, brain activity, and immune function during patients with anxiety states receiving TCM Daoyin intervention. Thus, the aims of the prospective randomized study are: (1) to examine the effects of TCM Daoyin training on reducing symptoms of anxiety, (2) to measure brain activity by using functional magnetic resonance imaging (fMRI), and (3) to assess Immune function.

DETAILED DESCRIPTION:
Anxiety is one of the most common mental health problems in the world. But there is a lack of sufficient no-drug intervention for relieving the anxious symptoms. The study focuses on mild and early anxiety disorder, which symptoms are not sufficiently severe, numerous, or persistent to justify a diagnosis of an anxiety disorder.

TCM Daoyin is a form of mind-body exercise with a profound philosophical foundation rooted in Chinese culture. Previous studies have provided some evidence of beneficial effects on TCM Daoyin for anxiety, such as Baduanjin and Liuzijue. However, the effects and neurophysiology mechanisms of TCM Daoyin on patients with anxiety state are yet to be further investigated.

This is a two-group prospective, randomized, assessor-blinded trial, planning to enroll 20 participants (10 for TCM Daoyin intervention group receiving health education plus a TCM Daoyin training program, and 10 for health education control group only receiving health education).

The aims of the prospective randomized study are: (1) to examine the effects of TCM Daoyin training on reducing symptoms of anxiety, (2) to measure brain activity by using functional magnetic resonance imaging (fMRI), and (3) to assess Immune function.

ELIGIBILITY:
Inclusion Criteria:

* Subject with a primary mental health complaint of anxiety.
* Anxiety 14≤HAMA-14≤29, Depression 7≤HAMD-17<14.
* Subject has no history of psychotropic medication or has been off medication for more than 6 months.
* Right-handed, aged 18 to 65, male or female.
* Subject has a clear mind and the ability to lead an independent life.
* Subject agrees to participate in fMRI scan and provide signed informed consent.

Exclusion Criteria:

* Subject with definite clinical diagnosis of anxiety disorder and depression disorder by ICD-10.
* Subject with bipolar disorder, psychotic disorder (e.g., schizophrenia), organic mental disorder (e.g., Alzheimer's disease).
* Subject with alcohol abuse, substance dependence and suicidal ideation in past-year, or currently taking psychiatric medication, or current serious suicidal attempt.
* Subject with serious current unstable medical illness.
* Subject has claustrophobia, or any contraindication unable or unwilling to participate in fMRI scan.
* Subject is clinically unable to participate in TCM Daoyin training program.
* Subject is pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
14-item Hamilton Anxiety Rating Scale | Change from Baseline HAMA-14 at 12 weeks
  The 14-item Hamilton Anxiety Rating Scale (HAMA-14) is a clinician-rated assessment (structured interview) of patients' anxious symptoms. Questions focus on anxious symptoms during the past 7 days, and higher cumulative scores indicate more severe anxiety.
  The HAMA-14 are rated on 5 grades ranging from 0(no symptom) to 4 (very severe). The total score ranges from 0 to 56. 29 or more on HAMA means severe anxiety disorders, 21 to 28 on HAMA means obvious anxiety disorders, 14 to 20 on HAMA means anxiety disorders, 8 to 13 on HAMA means suspicious anxiety disorders, 7 or less means no anxiety disorders.

SECONDARY OUTCOMES:
17-item Hamilton Depression Rating Scale | Change from Baseline HAMD-17 at 12 weeks
  The 17-item Hamilton Depression Rating Scale (HAMD-17) is a clinician-rated assessment (structured interview) of patients' depressive symptoms. Questions focus on depressive symptoms during the past 7 days, and higher cumulative scores indicate more severe depression.
  The HAMD-17 are rated on 5 grades ranging from 0(no symptom) to 4 (very severe). The total score ranges from 0 to 52. 25 or more on HAMD means severe depression disorders, 18 to 24 on HAMD means moderate depression, 13 to 17 on HAMD means mild depression disorders, 8 to 12 on HAMD means suspicious depression disorders, 7 or less means no depression disorders.
Depression, Anxiety and Stress Scale-21 item | Baseline
  The Depression, Anxiety and Stress Scale-21 item (DASS-21) is a self-rated assessment of patients' depressive, anxious and stress symptoms. Questions focus on depressive, anxious and stress symptoms during the past 7 days, and higher cumulative scores indicate more severe depression, anxiety and stress. Subscale scores are calculated as the sum of the responses to the seven items from each subscale multiplied by 2. The cutoffs for depression, anxiety, and stress are >9, >7, and >14, respectively.
Depression, Anxiety and Stress Scale-21 item | 6 weeks
  The Depression, Anxiety and Stress Scale-21 item (DASS-21) is a self-rated assessment of patients' depressive, anxious and stress symptoms. Questions focus on depressive, anxious and stress symptoms during the past 7 days, and higher cumulative scores indicate more severe depression, anxiety and stress. Subscale scores are calculated as the sum of the responses to the seven items from each subscale multiplied by 2. The cutoffs for depression, anxiety, and stress are >9, >7, and >14, respectively.
Depression, Anxiety and Stress Scale-21 item | 12 weeks
  The Depression, Anxiety and Stress Scale-21 item (DASS-21) is a self-rated assessment of patients' depressive, anxious and stress symptoms. Questions focus on depressive, anxious and stress symptoms during the past 7 days, and higher cumulative scores indicate more severe depression, anxiety and stress. Subscale scores are calculated as the sum of the responses to the seven items from each subscale multiplied by 2. The cutoffs for depression, anxiety, and stress are >9, >7, and >14, respectively.
Functional magnetic resonance imaging (fMRI) | Baseline
  The fMRI scans will be employed to assess whether engaging in TCM Daoyin training program does or does not alter structural imaging and functional imaging of brain activation. Changes in Blood Oxygen Level Dependent (BOLD) Response is investigated in resting state fMRI and task fMRI.
Functional magnetic resonance imaging (fMRI) | 12 weeks
  The fMRI scans will be employed to assess whether engaging in TCM Daoyin training program does or does not alter structural imaging and functional imaging of brain activation. Changes in Blood Oxygen Level Dependent (BOLD) Response is investigated in resting state fMRI and task fMRI.
Immune function | Change from Baseline immune function at 12 weeks
  CD3, CD4, CD8, IL-1β, IL-6 and TNF-α in blood samples will be measured to evaluate immune functions.
Adverse effects | 6 weeks
  During the intervention period, the doctors will ask specifically about, and record any adverse effect of the treatment that may have occurred.
Adverse effects | 12 weeks
  During the intervention period, the doctors will ask specifically about, and record any adverse effect of the treatment that may have occurred.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Qigong Research Institute, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No